CLINICAL TRIAL: NCT02600507
Title: Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Efficacy and Safety of ITI-007 Adjunctive to Lithium or Valproate in the Treatment of Patients With Major Depressive Episodes Associated With Bipolar I or Bipolar II Disorder
Brief Title: Clinical Trial Evaluating ITI-007 as an Adjunctive Therapy to Lithium or Valproate for the Treatment of Bipolar Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-007-402
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2021-04

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — lumateperone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lumateperone 28 mg (ITI-007 40 mg tosylate) (Experimental): Lumateperone 28 mg (ITI-007 40 mg tosylate) administered orally as capsules once daily for 6 weeks
  Interventions: Drug: Lumateperone (ITI-007)
- Lumateperone 42 mg (ITI-007 60 mg tosylate) (Experimental): Lumateperone 42 mg (ITI-007 60 mg tosylate) administered orally as capsules once daily for 6 weeks
  Interventions: Drug: Lumateperone (ITI-007)
- Placebo (Placebo Comparator): Placebo administered orally as visually-matched capsules once daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lumateperone (ITI-007)
  Arms: Lumateperone 28 mg (ITI-007 40 mg tosylate); Lumateperone 42 mg (ITI-007 60 mg tosylate)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy and safety of ITI-007 adjunctive to lithium or valproate in a randomized, double-blind, parallel-group, placebo-controlled, multi-center study in patients diagnosed with Bipolar I or Bipolar II disorder having a major depressive episode.

ELIGIBILITY:
Inclusion Criteria:

* male or female subjects of any race, ages 18-75 inclusive, with a clinical diagnosis of Bipolar I or Bipolar II disorder
* experiencing a current major depressive episode
* treatment with either lithium or valproate and inadequate therapeutic response of depressive symptoms

Exclusion Criteria:

* any subject unable to provide informed consent
* any female subject who is pregnant or breastfeeding
* any subject judged to be medically inappropriate for study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Kozauer, MD, Study Director — Intra-Cellular Therapies, Inc.
Locations (71):
- United States (42):
  - Clinical Site, Rogers, Arkansas
  - Clinical Site, Cerritos, California
  - Clinical Site, Costa Mesa, California
  - Clinical Site, Culver City, California
  - Clinical Site, Garden Grove, California
  - Clinical Site, Glendale, California
  - Clinical Site, Lemon Grove, California
  - Clinical Site, Oceanside, California
  - Clinical Site, Pico Rivera, California
  - Clinical Site, Riverside, California
  - Clinical Site, San Diego, California
  - Clinical Site, Santa Rosa, California
  - Clinical Site, Sherman Oaks, California
  - Clinical Site, Temecula, California
  - Clinical Site, Jacksonville, Florida
  - Clinical Site, Lauderhill, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Orange City, Florida
  - Clinical Site, Orlando, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Savannah, Georgia
  - Clinical Site, Chicago, Illinois
  - Clinical Site, Lake Charles, Louisiana
  - Clinical Site, Baltimore, Maryland
  - Clinical Site, O'Fallon, Missouri
  - Clinical Site, St Louis, Missouri
  - Clinical Site, Las Vegas, Nevada
  - Clinical Site, Berlin, New Jersey
  - Clinical Site, Cherry Hill, New Jersey
  - Clinical Site, Toms River, New Jersey
  - Clinical Site, Cedarhurst, New York
  - Clinical Site, New York, New York
  - Clinical Site, Rochester, New York
  - Clinical Site, Staten Island, New York
  - Clinical Site, Charlotte, North Carolina
  - Clinical Site, Cincinnati, Ohio
  - Clinical Site, Dayton, Ohio
  - Clinical Site, Garfield Heights, Ohio
  - Clinical Site, Allentown, Pennsylvania
  - Clinical Site, Philadelphia, Pennsylvania
  - Clinical Site, The Woodlands, Texas
  - Clinical Site, Everett, Washington
- Bulgaria (10):
  - Clinical Site, Burgas
  - Clinical Site, Kardzhali
  - Clinical Site, Lovech
  - Clinical Site, Pleven
  - Clinical Site, Plovdiv
  - Clinical Site, Rousse
  - Clinical Site, Sofia
  - Clinical Site, Varna
  - Clinical Site, Veliko Tarnovo
  - Clinical Site, Vratsa
- Russia (7):
  - Clinical Site, Moscow
  - Clinical Site, Nizhny Novgorod
  - Clinical Site, Omsk
  - Clinical Site, Saint Petersburg
  - Clinical Site, Samara
  - Clinical Site, Saratov
  - Clinical Site, Tomsk
- Serbia (4):
  - Clinical Site, Belgrade
  - Clinical Site, Kovin
  - Clinical Site, Novi Sad
  - Clinical Site, Šumadija
- Ukraine (8):
  - Clinical Site, Ivano-Frankivsk
  - Clinical Site, Kharkiv
  - Clinical Site, Kropyvnytskyi
  - Clinical Site, Odesa
  - Clinical Site, Poltava
  - Clinical Site, Smila
  - Clinical Site, Vasylkiv
  - Clinical Site, Vinnytsia

REFERENCES:
- [Derived] Suppes T, Durgam S, Kozauer SG, Chen R, Lakkis HD, Davis RE, Satlin A, Vanover KE, Mates S, McIntyre RS, Tohen M. Adjunctive lumateperone (ITI-007) in the treatment of bipolar depression: Results from a randomized placebo-controlled clinical trial. Bipolar Disord. 2023 Sep;25(6):478-488. doi: 10.1111/bdi.13310. Epub 2023 Feb 26. PMID 36779257

RESULTS

PARTICIPANT FLOW:
Groups:
- Lumateperone 28 mg (ITI-007 40 mg Tosylate): Lumateperone 28 mg (ITI-007 40 mg tosylate) administered orally as capsules once daily for 6 weeks
  Lumateperone 28 mg
- Lumateperone 42 mg (ITI-007 60 mg Tosylate): Lumateperone 42 mg (ITI-007 60 mg tosylate) administered orally as capsules once daily for 6 weeks
  Lumateperone 42
- Placebo: Placebo administered orally as visually-matched capsules once daily for 6 weeks
  Placebo
Period: Overall Study
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo
Started | 176 | 177 | 175 (176 patients were randomized to the placebo treatment group but only 175 patients took study drug. The number completed and discontinued is based on the 175 patients that took study drug.)
Completed | 147 | 133 | 150
Not Completed | 29 | 44 | 25
Not completed — Adverse Event | 3 | 15 | 5
Not completed — Lack of Efficacy | 3 | 8 | 5
Not completed — Lost to Follow-up | 3 | 5 | 2
Not completed — Protocol Violation | 12 | 4 | 4
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 11 | 7
Not completed — Other | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lumateperone 42 mg (ITI-007 60 mg Tosylate): Lumateperone 42 mg (ITI-007 60 mg tosylate) administered orally as capsules once daily for 6 weeks
  Lumateperone 42 mg
- Total: Total of all reporting groups
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo | Total
Number analyzed (Participants) | 176 | 177 | 175 | 528
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (13.56) | 44.7 (12.60) | 45.1 (12.93) | 44.6 (13.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 109 | 98 | 308
  Male | 75 | 68 | 77 | 220
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 153 | 156 | 157 | 466
  Black or African American | 22 | 20 | 14 | 56
  Asian | 0 | 0 | 3 | 3
  Other | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 59 | 58 | 56 | 173
  Ukraine | 21 | 21 | 15 | 57
  Bulgaria | 49 | 45 | 48 | 142
  Serbia | 16 | 16 | 20 | 52
  Russia | 31 | 37 | 36 | 104
Montgomery-Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — The Montgomery-Asberg Depression Rating Scale (MADRS) is a clinician-rated 10 item scale to assess depressive symptoms. Each item is rated on a 7-point scale from 0-6. The total score ranges from 0 to 60 with a higher score indicating increased severity of depressive symptoms.
  units on a scale | 32.5 (5.55) | 32.3 (4.96) | 32.2 (5.23) | 32.3 (5.24)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician-rated 10 item scale to assess depressive symptoms. Each item is rated on a 7-point scale from 0-6. The total score ranges from 0 to 60 with a higher score indicating increased severity of depressive symptoms.
Time Frame: Baseline to Day 43
Population: Intent-to-Treat (ITT) Set contains all randomized patients who received at least one dose of study medication and had a valid baseline (pre-dose) measurement and at least one valid post-baseline measurement of MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo
Number analyzed (Participants) | 171 | 174 | 174
score on a scale | -16.2 (0.79) | -16.9 (0.81) | -14.5 (0.79)
Statistical Analysis 1: Comparison: Lumateperone 42 mg (ITI-007 60 mg Tosylate) vs Placebo; Test type: Superiority; p = 0.021, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -2.4, 95% CI 2-sided [-4.42 to -0.37], Standard Error of Mean 1.03
Statistical Analysis 2: Comparison: Lumateperone 28 mg (ITI-007 40 mg Tosylate) vs Placebo; Test type: Superiority; p = 0.099, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -1.7, 95% CI 2-sided [-3.65 to 0.32], Standard Error of Mean 1.01

2. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale-Bipolar Version-Severity (CGI-BP-S) Depression Score
Description: The Clinical Global Impression Scale-Bipolar Version-Severity (CGI-BP-S) Depression Score is a clinician-rated scale that measures the patient's current state of depression from 1 (not ill at all) to 7 (among the most extremely ill).
Time Frame: Baseline to Day 43
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo
Number analyzed (Participants) | 171 | 174 | 174
score on a scale | -1.7 (0.09) | -1.8 (0.10) | -1.5 (0.09)
Statistical Analysis 1: Comparison: Lumateperone 42 mg (ITI-007 60 mg Tosylate) vs Placebo; Test type: Superiority; p = 0.008, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-0.59 to -0.09], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Lumateperone 28 mg (ITI-007 40 mg Tosylate) vs Placebo; Test type: Superiority; p = 0.040, Mixed Effects Model for Repeated Measure; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-0.50 to -0.01], Standard Error of Mean 0.12

ADVERSE EVENTS:
Time Frame: From signing ICF until end of study procedures (~10 weeks), including 6 weeks of double-blind treatment.
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/177 | 0/175
Serious Adverse Events (participants affected / at risk) | 0/176 | 1/177 | 0/175
Other Adverse Events (participants affected / at risk) | 50/176 | 47/177 | 28/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lumateperone 28 mg (ITI-007 40 mg Tosylate) (N=176) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) (N=177) | Placebo (N=175)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lumateperone 28 mg (ITI-007 40 mg Tosylate) (N=176) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) (N=177) | Placebo (N=175)
Headache (Nervous system disorders) | 23 | 20 | 20
Somnolence (Nervous system disorders) | 13 | 20 | 6
Dizziness (Nervous system disorders) | 18 | 19 | 4
Nausea (Gastrointestinal disorders) | 10 | 15 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/07/NCT02600507/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT02600507/SAP_001.pdf